CLINICAL TRIAL: NCT01820546
Title: Flow Cytometric Definition and Prognostic Effects of Multiple Myeloma Cancer Stem Cells
Brief Title: Cancer Stem Cells in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Mehmet Ozen, MD, Ankara University
Other Study IDs: TR06
Record Dates: First submitted 2013-03-26; First posted 2013-03-28 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow
Oversight: Data Monitoring Committee: No

SUMMARY:
In multiple myeloma "cancer stem" cells can be defined and quantified with flow cytometry. More, these cells can be related to treatment response.

DETAILED DESCRIPTION:
The investigators' hypothesis is that, multiple myeloma plasma cells derivate from principal cells that is called "cancer or progenitor stem cell". In multiple myeloma to define immunophenotyping features of these "cancer stem cells" with flow cytometry and to show their prognostic value and check for any relationship between cancer stem cell quantification and chemotherapy response are main aims of this study.

ELIGIBILITY:
Inclusion Criteria:

* New Diagnosed or Relapsed Multiple Myeloma
* Routine Bone Marrow Aspiration will be done

Exclusion Criteria:

* Bone Marrow Aspiration is not Needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New Diagnosed or Relapsed Multiple Myeloma Patients
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Treatment Response | 3 months
  After 3 courses chemotherapy treatment response

SECONDARY OUTCOMES:
Treatment Response | 6 months
  After 6 courses chemotherapy treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozen, MD, Principal Investigator
Locations (1):
- Ankara University Hematology Unit, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Matsui W, Huff CA, Wang Q, Malehorn MT, Barber J, Tanhehco Y, Smith BD, Civin CI, Jones RJ. Characterization of clonogenic multiple myeloma cells. Blood. 2004 Mar 15;103(6):2332-6. doi: 10.1182/blood-2003-09-3064. Epub 2003 Nov 20. PMID 14630803